CLINICAL TRIAL: NCT04539548
Title: A Randomized, Parallel-Arm, Active Control, Multi-Center Study Assessing the Safety And Efficacy Of Dextenza® for the Treatment Of Ocular Pain and Inflammation Following Surgery for Pediatric Cataract
Brief Title: A Study Assessing the Safety and Efficacy of Dextenza® for the Treatment of Ocular Pain and Inflammation Following Surgery for Pediatric Cataract
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLN-Protocol-0050
Record Dates: First submitted 2020-08-27; First posted 2020-09-07 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Cataract
Keywords: Dextenza, dexamethasone ophthalmic insert
MeSH Terms: conditions — Cataract | interventions — Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dextenza (Experimental): 1 dosing group - 37 eyes treated with Dextenza
  Interventions: Drug: Dextenza Ophthalmic Insert
- Prednisolone (Active Comparator): 1 dosing group - 32 eyes treated with Prednisolone
  Interventions: Drug: Prednisolone acetate ophthalmic suspension USP 1%

INTERVENTIONS:
Drug: Dextenza Ophthalmic Insert — 0.4mg insert for intracanalicular use
  Other Names: DEXTENZA
  Arms: Dextenza
Drug: Prednisolone acetate ophthalmic suspension USP 1% — 1 drop at end of surgery, followed by:
  1 drop 4 x QID for one week.
  1 drop 3 x QID for one week.
  1 drop BID for one week.
  1 drop QD for one week
  Arms: Prednisolone

SUMMARY:
To assess the safety of Dextenza compared to an active control, prednisolone acetate suspension, for the treatment of postoperative pain and inflammation following ocular surgery for pediatric cataract.

DETAILED DESCRIPTION:
Randomized, parallel-arm, active control, multi-center study assessing the safety of Dextenza for the treatment of ocular pain and inflammation following surgery for pediatric cataract. The subjects will be followed for approximately 2-3 months from screening to the last visit.

ELIGIBILITY:
Inclusion Criteria:

* Is 0-5 years of age (up to the day before the subject turns 6 years of age). In the event that a subject aged 0-5 years enrolls in the study and then undergoes a second cataract surgery in the contralateral eye during the study period, the subject remains eligible for participation for both eyes, regardless if the second surgery occurs when the subject is >5 years of age)
* Has a cataract and is expected to undergo primary cataract surgery with or without implantation of a posterior chamber intraocular lens

Exclusion Criteria:

* Any intraocular inflammation in the study eye present during the screening slit lamp examination
* Has ocular hypertension (defined as IOP of >21 mmHg), or glaucoma or is on medications to treat ocular hypertension or glaucoma or has a history of IOP spikes in either eye including steroid-related IOP increases
* Evidence of acute external ocular infections (bacterial, viral and/or fungal such as vaccinia, varicella, and other viral diseases of the cornea and conjunctiva), tuberculosis of the eye; corneal dystrophies; active corneal ulcers, intraocular infections, dysthyroid ophthalmopathy, active chalazion, or uncontrolled blepharitis in the study eye

Ages: 0 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to approximately 42 days after surgery
  Number of Ocular Treatment Emergent Adverse Events (TEAEs) and Non-ocular Treatment Emergent Adverse Events (TEAEs)
Subject FLACC Pain Assessment | From screening through day 42
  Behavioral Observation Pain Rating Scale from 0 (no pain) to 10 (most pain).
IOP | From screening, then day 2 through 42
  IOP measured in units of mmHg.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Ocular Therapeutix, Aurora, Colorado
  - Ocular Therapeutix, Fort Collins, Colorado
  - Ocular Therapeutix, Jacksonville, Florida
  - Ocular Therapeutix, Indianapolis, Indiana
  - Ocular Therapeutix, Lexington, Kentucky
  - Ocular Therapeutix, Boston, Massachusetts
  - Ocular Therapeutix, Minneapolis, Minnesota
  - Ocular Therapeutix, Rochester, Minnesota
  - Ocular Therapeutix, St Louis, Missouri
  - Ocular Therapeutix, Erie, Pennsylvania
  - Ocular Therapeutix, Charleston, South Carolina
  - Ocular Therapeutix, Nashville, Tennessee
  - Ocular Therapeutix, Virginia Beach, Virginia
  - Ocular Therapeutix, Madison, Wisconsin